CLINICAL TRIAL: NCT07315451
Title: Comparison of Lateral Decubitus and Upright Sitting Positions in Measuring Intervertebral Space Via Ultrasound in Obese Volunteers
Status: Enrolling by invitation | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Emre Sanci, M.D., Asst. Prof., Kocaeli City Hospital
Other Study IDs: 2021-120
Record Dates: First submitted 2025-03-02; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Spinal Column; Lumbar Puncture; Ultrasonography; Position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to compare the lateral decubitus and upright sitting positions in determining the intervertebral space measured by ultrasound in participants whose body mass index was greater than 30 and older than eighteen years old. Additionally, comparison of the sagittal and long-axis paramedian oblique planes in determining the intervertebral space measured by ultrasound in this group of volunteers. Furthermore, assesment of the reliability of measurements performed by practitioners with varying levels of ultrasound experience.

DETAILED DESCRIPTION:
The study will be conducted in the Emergency Medicine Clinic of University of Health Sciences Kocaeli City Hospital. Participants over the age of 18 with a body mass index (BMI) of 30 or higher presenting to the emergency department will be included. After providing verbal information about the study, written informed consent will be obtained from participants who agree to take part. Participants will be evaluated by attending physicians in the emergency department, who will then inform the study investigators.

The upright sitting position is defined as the patient sitting upright on the stretcher with their legs hanging down the side, feet not touching the ground, and arms extended forward for support. The lateral decubitus position is defined as the patient lying on their side with their shoulders and hips perpendicular to the stretcher, knees flexed, and pulled toward the chest.

The ultrasound applications will be performed by two study investigators: one emergency medicine specialist with advanced ultrasound training and one with basic ultrasound training. Measurements will be taken first in the participant's preferred position (upright sitting or lateral decubitus) and then in the alternate position.

Since the traditional method for identifying the lumbar puncture (LP) site-known as Tuffier's line (the midpoint of the line connecting both anterior superior iliac spines in the lumbar region)-can be misleading in obese patients, the application site will be determined via ultrasound. An Esaote MyLab™ Gamma ultrasound device will be used, with the Esaote SL1543 linear probe as the first choice. If the linear probe does not provide adequate depth due to obesity, the Esaote SP2730 curved probe will be used.

For ultrasound application, the probe will initially be placed transversely just above the intragluteal fold, with the indicator pointing to the patient's left shoulder. Once the midline is identified, measurements will be performed in two planes: sagittal and long-axis paramedian oblique.

For the sagittal plane, the probe will be rotated 90 degrees with the indicator pointing toward the patient's head.

For the long-axis paramedian oblique plane, the probe will also be rotated 90 degrees toward the head but moved 1-2 cm laterally from the midline and angled slightly medially.

The probe will then be moved superiorly until the L4-L5 interspinal space is identified. The intervertebral space is defined as the hypoechoic region between hyperechoic spinous processes. Measurements will be taken from the L4-L5 and L3-L4 intervertebral spaces.

Each practitioner's measurements will include the distance to the ligamentum flavum, as well as data on whether the patient has undergone lumbar surgery, and their weight and height. These will be recorded in a pre-prepared standard data form. Practitioners will be blinded to each other's measurements to maintain objectivity.

ELIGIBILITY:
Inclusion Criteria:

* participants whose body mass index was greater than 30
* participants older than eighteen years old.

Exclusion Criteria:

* participants who have a history of lumbar surgery
* participants who have an infection on the lombar region
* pregnant volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who want to participate in the study will be included.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Lateral Decubitus and Upright Sitting Positions in Ultrasound Measurement of Intervertebral Space in Adults with a BMI Over 30 | Baseline
  The primary outcome of the study is to compare the lateral decubitus and upright sitting positions in determining the intervertebral space measured by ultrasound in participants whose body mass index was greater than 30

SECONDARY OUTCOMES:
Comparison of Sagittal and Paramedian Oblique Planes for Ultrasound Measurement of Intervertebral Space | Baseline
  The secondary outcome measure was comparison of the sagittal and long-axis paramedian oblique planes in determining the intervertebral space measured by ultrasound in participants whose body mass index was greater than 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roberts and Hedges' Clinical Procedures in Emergency Medicine and Acute Care. Editors: Roberts, J. R., Custalow, C. B., & Thomsen, T. W. . Seventh edition. Philadelphia, PA: Elsevier
- [Background] Nomura JT, Leech SJ, Shenbagamurthi S, Sierzenski PR, O'Connor RE, Bollinger M, Humphrey M, Gukhool JA. A randomized controlled trial of ultrasound-assisted lumbar puncture. J Ultrasound Med. 2007 Oct;26(10):1341-8. doi: 10.7863/jum.2007.26.10.1341. PMID 17901137
- [Background] Ferre RM, Sweeney TW. Emergency physicians can easily obtain ultrasound images of anatomical landmarks relevant to lumbar puncture. Am J Emerg Med. 2007 Mar;25(3):291-6. doi: 10.1016/j.ajem.2006.08.013. PMID 17349903
- [Background] Stiffler KA, Jwayyed S, Wilber ST, Robinson A. The use of ultrasound to identify pertinent landmarks for lumbar puncture. Am J Emerg Med. 2007 Mar;25(3):331-4. doi: 10.1016/j.ajem.2006.07.010. PMID 17349909
- [Background] Huang MY, Lin AP, Chang WH. Ultrasound-assisted localization for lumbar puncture in the ED. Am J Emerg Med. 2008 Oct;26(8):955-7. doi: 10.1016/j.ajem.2008.03.007. No abstract available. PMID 18926360
- [Background] Furness G, Reilly MP, Kuchi S. An evaluation of ultrasound imaging for identification of lumbar intervertebral level. Anaesthesia. 2002 Mar;57(3):277-80. doi: 10.1046/j.1365-2044.2002.2403_4.x. PMID 11892638
- [Background] Shi D, Perice L, Grimaldi C, Perera T, Nelson M. Ultrasound Measurement of the Intervertebral Space in the Lateral Recumbent Versus Sitting Positions. J Emerg Med. 2021 Dec;61(6):705-710. doi: 10.1016/j.jemermed.2021.07.015. Epub 2021 Aug 29. PMID 34465511
- [Background] Andreas Dewitz, Robert A. Jones, Jessica G. Resnick, and Michael B. Stone. Additional Ultrasound-Guided Procedures. Ma and Mateer's Emergency Ultrasound. Editors: O John Ma; James R Mateer; Robert F Reardon; Scott Joing. Third Edition. New York : McGraw-Hill Education. 2014.